CLINICAL TRIAL: NCT00708695
Title: Age-17 Follow-up of Home Visiting Intervention
Acronym: MemphisY17
Status: Completed | Type: Observational
Sponsor: University of Colorado, Denver (Other)
Collaborators: University of Rochester (Other); Emory University (Other); University of Colorado, Boulder (Other); RTI International (Other); National Institute on Drug Abuse (NIDA) (NIH); Yale University (Other)
Responsible Party: Sponsor
Other Study IDs: 08-0616; R01DA021624 (NIH)
Record Dates: First submitted 2008-05-27; First posted 2008-07-02 (Estimated); Last update posted 2022-05-04 (Actual); Status verified 2022-04

CONDITIONS: Antisocial Behavior; Psychopathology; Substance Use; HIV Infections
Keywords: nurse; home visits; pregnancy; welfare; child development; Child Rearing; Reproductive Behavior; Risk Reduction Behavior
MeSH Terms: conditions — Antisocial Personality Disorder; Substance-Related Disorders; HIV Infections; Reproductive Behavior; Risk Reduction Behavior | interventions — Nurses, Community Health

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Spit samples will be taken.
Oversight: Data Monitoring Committee: Yes

GROUPS / COHORTS (2):
- Treatment 2: Transportation, Child Screening/Referral: The 514 families received: 1) free transportation for prenatal care; and 2) child developmental screening and referral services.
- Treatment 4: Nurse Home Visiting through Age 2: The 228 families: 1) free transportation for prenatal care; 2) nurse home-visiting during pregnancy and through child's second birthday; and 3) child developmental screening and referral.
  Interventions: Behavioral: Nurse Home Visiting

INTERVENTIONS:
Behavioral: Nurse Home Visiting — Visits from nurses from mid-pregnancy to child age 2 years.
  Groups: Treatment 4: Nurse Home Visiting through Age 2

SUMMARY:
This study is a longitudinal follow-up of 670 primarily African-American women and their 17-year-old firstborn children enrolled since 1990 in a highly significant randomized controlled trial (RCT) of prenatal and infancy home visiting by nurses. Nurses in this program are charged with improving pregnancy outcomes, child health and development, and maternal economic self-sufficiency. This follow-up examines whether earlier program effects on maternal and child functioning lead to less violent antisocial behavior, psychopathology, substance use and use-disorders, and risk for HIV; whether these effects are greater for those at both genetic and environmental risk; and whether program effects replicate those found with whites in an earlier trial.

DETAILED DESCRIPTION:
This study is a longitudinal follow-up of 670 primarily African-American women and their 18-year-old firstborn children enrolled since 1990 in a randomized controlled trial (RCT) of prenatal and infancy home visiting by nurses. Nurses in this program are charged with improving pregnancy outcomes, child health and development, and maternal economic self-sufficiency.1 This follow-up examines whether earlier program effects on maternal and child functioning 2-7 lead to less violent antisocial behavior, psychopathology, substance use and use-disorders, and risk for HIV; whether these effects are greater for those who carry genetic susceptibility to the environment and are at environmental risk; and whether program effects replicate those found with whites in an earlier trial.8-10 Results from earlier phases of follow-up from this trial found that the Memphis program affected women's prenatal health, fertility, partner relations, and use of welfare; children's injuries, cognition, language, achievement, conduct, depression/anxiety, and use of substances through child age 12.2-7 Program effects on maternal life-course were concentrated among mothers with higher psychological resources (better intellectual functioning, mental health, and sense of mastery), probably because higher-resource mothers could envision their success in the world of work, leading to better pregnancy planning and employment. Program effects on children were greater for those born to mothers with low psychological resources, because without help, low-resource mothers are especially challenged in the care of their children and their children function less well. Given the damaging effects of early stressors on developing neural circuitry, and given that many early neural developmental insults do not become fully evident until synaptic pruning is complete in late adolescence and early adulthood, there was reason to expect this early intervention would have enduring effects at youth age 18.

Hypotheses for Primary Grant

We specified hypotheses based upon the pattern of results found through child age 12, and separated them into primary and secondary hypotheses. Following the original formulation of hypotheses, we edited them to take into account results from the earlier Elmira trial10 that were analyzed following the submission of the proposal for the current phase of follow-up in Memphis. We had originally hypothesized that program effects would be more pronounced for mothers and children living in the most disadvantaged neighborhoods in Memphis, but realized as these data were being gathered that virtually all of the participants in the Memphis trial lived in neighborhoods that were so disadvantaged that there was little meaningful variation among neighborhoods, and therefore removed this aspect of our hypotheses. We also found that it was impossible to consistently gather information from children's school records on outcomes like conduct grades from hundreds of schools, so substituted high school graduation as a secondary outcome. These refined hypotheses were specified prior to the completion of data gathering and any analysis of treatment-control differences. We specify the original hypotheses and then indicate the revised hypotheses for maternal and child outcomes. Compared to control-group counterparts:

Original Maternal Outcomes Hypotheses

1. (Primary) The program will continue to improve maternal life-course (fewer short inter-birth intervals, less use of welfare, more stable partner relations), especially for mothers with higher psychological resources.
2. (Secondary) The program will reduce maternal substance use disorders (SUDs) and depression, effects that will be more pronounced for a) mothers with low psychological resources, and b) those living in the most disadvantaged neighborhoods at registration.

Revised Maternal Outcome Hypotheses

1. (Primary) The program will continue to improve maternal life-course (reflected in total costs of welfare - SNAP, TANF, Medicaid), especially for mothers with higher psychological resources.
2. (Secondary) The program will reduce maternal substance use disorders (SUDs) and depression.

   Original Child Outcomes Hypotheses
3. (Primary) The program will improve the health and development of firstborn children who will exhibit: a) superior cognitive, language, and academic functioning, and executive cognitive functioning (ECF); b) less depression and anxiety; c) fewer failed conduct grades and school disciplinary actions, d) less violent behavior and gang membership, and fewer arrests, juvenile detentions, and convictions - especially for crimes involving interpersonal violence.
4. (Primary) The program will reduce youth risk for HIV infection, including a) use of substances and SUDs; b) risky sexual behaviors; c) sexually transmitted infections (STIs) and d) pregnancies.
5. (Primary) Program effects on youth will be more pronounced for a) males, b) those born to low-resource mothers, and c) those living in the most disadvantaged neighborhoods at registration.

Revised Child Outcome Hypotheses 3. (Primary) The program will improve the health and development of firstborn children who will exhibit: a) superior cognitive, language, and academic functioning; b) less depression and anxiety; d) less gang membership, and fewer arrests, convictions, and self-reported antisocial behavior - especially for crimes involving interpersonal violence.

4. (Primary) The program will reduce youth risk for HIV infection, pregnancies, births, use of substances, and SUDs.

5. (Secondary) The program will improve firstborn children's executive cognitive functioning (ECF); and rates of high school graduation.

6. (Primary) Program effects on cognitive, language, and academic functioning, and executive cognitive functioning will be more pronounced among those born to low-resource mothers and on arrests and convictions among females.

Maternal and Child Outcomes (Not Revised) 7. (Secondary) Program effects on mothers and youth, in preliminary analyses, will be more pronounced for those with genetic vulnerabilities:

1. Effects on youth depression and anxiety will be greater for those with low-activity genotypes (S/S, LG/LG, S/LG) of the serotonin transporter gene (SLC6A4) promoter polymorphism, 5-HTTLPR, compared to those with high-activity genotypes (LA/LA); effects on these outcomes will be of intermediate magnitude for those with intermediate activity-level genotypes (S/LA, LA/LG).
2. Effects on youth violent antisocial behavior, SUDs, and risky sexual behavior will be more pronounced among males with the MAOA-LPR low activity alleles compared to males with MAOA-LPR high activity alleles, and among both males and females with 2 copies of the high-activity Val allele of the COMT Val158Met polymorphism compared to those with 2 copies of the low-activity met allele or heterozygotes.
3. Effects on maternal SUDs will be concentrated among mothers with 2 copies of the Val158 alleles.
4. Effects on child outcomes will be more pronounced among youth born to mothers with either 1) the S/S, S/LG and "LG/LG" (low-activity) genotypes of 5-HTTLPR (conferring susceptibility for depression under adversity) or 2) 2 copies of the high activity COMT Val158 allele (conferring susceptibility to compromised ECF and SUDs under conditions of adversity).

   8. (Secondary) Program effects on adolescent functioning will be explained by its improvement in prenatal health, early care of the child, maternal life-course, and earlier child academic and behavioral functioning.

   Examination of Intervention Effects on Subsequent Children With an administrative supplement, we addressed the following questions focused on subsequent children born within 5 years of the first child. Note that these questions were framed with no specific hypotheses about the degree to which particular subgroups would benefit from the intervention, given that intervention impact on pregnancy planning had been most pronounced on women with higher psychological resources.
   1. To what degree does this program improve the health and development of subsequent children in terms of their a) language, academic, and executive cognitive functioning (ECF); b) depression and anxiety; c) failed conduct grades, d) violent behavior and gang membership, and e) arrests, juvenile detentions, and convictions, especially for violent crimes?
   2. To what degree does this program reduce subsequent children's risk for HIV infection, including a) use and abuse of substances; b) risky sexual behaviors; c) sexually transmitted infections (STIs) and d) pregnancies?
   3. To what degree are the program effects on subsequent children more pronounced for a) males, b) those born to high-resource mothers, and c) those living in the most disadvantaged neighborhoods at registration?
   4. To what degree are program effects on subsequent children's functioning explained by its earlier impact on a) the timing and rates of subsequent births; b) families' use of welfare-related services; c) stability in partner relationships; d) improvements in neighborhood contexts; and e) antisocial behavior among the first-borns?

   Aims of the Benefit-Cost Analysis

   With an administrative supplement, we conducted a benefit-cost analysis of NFP in Memphis. The benefit-cost study was designed to:
   1. Estimate return on investment in Memphis NFP from the perspectives of government, society and individual participants.
   2. Estimate the quality-adjusted life year (QALY) savings produced by the Memphis NFP.
   3. Combine effectiveness estimates from Memphis NFP with those from other NFP evaluations and produce a combined estimate.
   4. Develop a model that states can use to estimate the value of funding NFP programs.
   5. Compare the cost-effectiveness of the NFP to other commonly delivered childhood interventions.

ELIGIBILITY:
Inclusion Criteria:

* Women who were enrolled in the New Mothers Study and their children as described in Study Population Description.

Exclusion Criteria:

* Women who were not enrolled in the New Mothers Study and their children as described in the Study Population Description.

Ages: 17 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Very low-income African-Americans living in a major urban area. In this trial, 1,138 low-income pregnant women (98% unmarried, 67% <19 years old, 92% African-American) were randomly assigned to experimental or comparison services; 742 were followed after delivery. The sample resided in extraordinarily stressful neighborhoods and endured extreme poverty. At registration, 85% of the sample had incomes below the federal poverty guidelines.
Sampling Method: Probability Sample
Enrollment: 1880 (Actual)
Dates: Start 2008-05; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Maternal life-course (reflected in reduced total public benefit expenditures for SNAP, AFDC/TANF, and Medicaid). | through first child age 18
  Public benefit expenditures estimated from review of state administrative records and maternal report of all children's birth dates. Program effects on public-benefit expenditures hypothesized to be especially pronounced for mothers with higher psychological resources.
Cognitive, language, and academic functioning among first-born children. | at youth age 18
  Direct tests of youth cognitive, language, and academic functioning. Program effects in this domain hypothesized to be most pronounced for children born to mothers with low psychological resources.
Youth depression and anxiety | at youth age 18
  Measure of internalizing disorders based upon youth self-report.
Youth gang membership, arrests, convictions, and self-reported antisocial behavior, especially for crimes involving interpersonal violence. | at youth age 18
  Self-reported involvement with criminal justice system and antisocial behavior. Program effects on arrests and convictions hypothesized to be greater for females.
Youth risk for HIV infection, pregnancies, births, use of substances, and SUDs. | at youth age 18.
  Outcomes based upon self-report and urine assays for STI's and substance use.

SECONDARY OUTCOMES:
Reduced maternal substance use disorders (SUDs) and depression. | at youth age 18
  Based upon maternal self-report of SUDs and depression.
Improved child executive cognitive functioning, and rates of high school graduation. | at youth age 18
  Based upon direct tests of risky decision making, impulsivity, facial recognition, verbal working memory) and records of high school graduation. Program effects in this domain hypothesized to be more pronounced for children born to mothers with low psychological resources.

OTHER OUTCOMES:
Cumulative subsequent pregnancies - mothers | through youth age 18
  Self-reported number of subsequent pregnancies, pregnancy outcomes, live births, low-birth weight newborns, and birth dates. Program effects on cumulative pregnancies and births hypothesized to be more pronounced among mothers with high psychological resources.
Pregnancies - youth | through youth age 18
  Self-reported pregnancies and pregnancy outcomes.
Relationship with Current Partner | at youth age 18
  Self-reported duration and quality of relationship, cohabitation, marriage, partner employment, and relationship to first-born child

CONTACTS AND LOCATIONS:
Overall Officials: David L Olds, PhD, Principal Investigator — University of Colorado, Denver
Locations (1):
- Memphis Study Office, Memphis, Tennessee, United States

IPD SHARING:
Plan to Share IPD: Yes
Deidentified individual participant data (including data dictionaries) will be made available in addition to study protocols, the statistical analysis plan, and the informed consent form. The data will be made available on publication to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: 2 years, beginning December 31st, 2023
Access Criteria: The data will be made available on publication to researchers who provide a methodologically sound proposal for use in achieving the goals of the approved proposal. Please contact Michael Knudtson, the study biostatistician, at michael.knudtson@cuanschutz.edu or 303-724-3199 for additional details.

REFERENCES:
- [Background] Kitzman H, Olds DL, Henderson CR Jr, Hanks C, Cole R, Tatelbaum R, McConnochie KM, Sidora K, Luckey DW, Shaver D, Engelhardt K, James D, Barnard K. Effect of prenatal and infancy home visitation by nurses on pregnancy outcomes, childhood injuries, and repeated childbearing. A randomized controlled trial. JAMA. 1997 Aug 27;278(8):644-52. PMID 9272896
- [Background] Kitzman H, Olds DL, Sidora K, Henderson CR Jr, Hanks C, Cole R, Luckey DW, Bondy J, Cole K, Glazner J. Enduring effects of nurse home visitation on maternal life course: a 3-year follow-up of a randomized trial. JAMA. 2000 Apr 19;283(15):1983-9. doi: 10.1001/jama.283.15.1983. PMID 10789666
- [Background] Olds DL, Kitzman H, Cole R, Robinson J, Sidora K, Luckey DW, Henderson CR Jr, Hanks C, Bondy J, Holmberg J. Effects of nurse home-visiting on maternal life course and child development: age 6 follow-up results of a randomized trial. Pediatrics. 2004 Dec;114(6):1550-9. doi: 10.1542/peds.2004-0962. PMID 15574614
- [Background] Olds DL, Kitzman H, Hanks C, Cole R, Anson E, Sidora-Arcoleo K, Luckey DW, Henderson CR Jr, Holmberg J, Tutt RA, Stevenson AJ, Bondy J. Effects of nurse home visiting on maternal and child functioning: age-9 follow-up of a randomized trial. Pediatrics. 2007 Oct;120(4):e832-45. doi: 10.1542/peds.2006-2111. PMID 17908740
- [Background] Olds DL, Kitzman HJ, Cole RE, Hanks CA, Arcoleo KJ, Anson EA, Luckey DW, Knudtson MD, Henderson CR Jr, Bondy J, Stevenson AJ. Enduring effects of prenatal and infancy home visiting by nurses on maternal life course and government spending: follow-up of a randomized trial among children at age 12 years. Arch Pediatr Adolesc Med. 2010 May;164(5):419-24. doi: 10.1001/archpediatrics.2010.49. PMID 20439792
- [Background] Kitzman HJ, Olds DL, Cole RE, Hanks CA, Anson EA, Arcoleo KJ, Luckey DW, Knudtson MD, Henderson CR Jr, Holmberg JR. Enduring effects of prenatal and infancy home visiting by nurses on children: follow-up of a randomized trial among children at age 12 years. Arch Pediatr Adolesc Med. 2010 May;164(5):412-8. doi: 10.1001/archpediatrics.2010.76. PMID 20439791
- [Background] Olds DL, Kitzman H, Knudtson MD, Anson E, Smith JA, Cole R. Effect of home visiting by nurses on maternal and child mortality: results of a 2-decade follow-up of a randomized clinical trial. JAMA Pediatr. 2014 Sep;168(9):800-6. doi: 10.1001/jamapediatrics.2014.472. PMID 25003802
- [Derived] Conti G, Smith J, Anson E, Groth S, Knudtson M, Salvati A, Olds D. Early Home Visits and Health Outcomes in Low-Income Mothers and Offspring: 18-Year Follow-Up of a Randomized Clinical Trial. JAMA Netw Open. 2024 Jan 2;7(1):e2351752. doi: 10.1001/jamanetworkopen.2023.51752. PMID 38236602
- [Derived] Kitzman H, Olds DL, Knudtson MD, Cole R, Anson E, Smith JA, Fishbein D, DiClemente R, Wingood G, Caliendo AM, Hopfer C, Miller T, Conti G. Prenatal and Infancy Nurse Home Visiting and 18-Year Outcomes of a Randomized Trial. Pediatrics. 2019 Dec;144(6):e20183876. doi: 10.1542/peds.2018-3876. Epub 2019 Nov 20. PMID 31748254
- [Derived] Olds DL, Kitzman H, Anson E, Smith JA, Knudtson MD, Miller T, Cole R, Hopfer C, Conti G. Prenatal and Infancy Nurse Home Visiting Effects on Mothers: 18-Year Follow-up of a Randomized Trial. Pediatrics. 2019 Dec;144(6):e20183889. doi: 10.1542/peds.2018-3889. Epub 2019 Nov 20. PMID 31748253
- [Derived] Enoch MA, Kitzman H, Smith JA, Anson E, Hodgkinson CA, Goldman D, Olds DL. A Prospective Cohort Study of Influences on Externalizing Behaviors Across Childhood: Results From a Nurse Home Visiting Randomized Controlled Trial. J Am Acad Child Adolesc Psychiatry. 2016 May;55(5):376-82. doi: 10.1016/j.jaac.2016.02.007. Epub 2016 Mar 2. PMID 27126851
- See also: Related Info — https://www.nursefamilypartnership.org/

DOCUMENTS (1):
  • Informed Consent Form (2018-03-16): https://cdn.clinicaltrials.gov/large-docs/95/NCT00708695/ICF_001.pdf